CLINICAL TRIAL: NCT00637676
Title: Randomized Trial of Tunneled Pleural Catheter Versus Standard Chest Tube in Management of Malignant Pleural Effusion in Patients With Partial Entrapment of the Lung
Brief Title: Tunneled Pleural Catheter in Partially Entrapped Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Head, Heidelberg University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2802
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Malignant Pleural Effusion
Keywords: malignant pleural effusion; subcutaneous tunneled drainage; talc pleurodesis
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Implantation of PleurX-Pleural catheter plus talc pleurodesis
  Interventions: Procedure: VATS, Talc-Pleurodesis, tunneled pleural drainage
- 2 (Active Comparator): talc pleurodesis, no implantation of PleurX-Pleural catheter
  Interventions: Procedure: VATS, Talc-pleurodesis

INTERVENTIONS:
Procedure: VATS, Talc-Pleurodesis, tunneled pleural drainage — poudrage of 4 gr talc into the pleural cavity implantation of tunneled pleural catheter
  Other Names: Device: PleurX-Pleural Catheter
  Arms: 1
Procedure: VATS, Talc-pleurodesis — poudrage of 4 gr. talc into the pleural cavity no tunneled pleural catheter
  Other Names: no PleurX-Pleural Catheter
  Arms: 2

SUMMARY:
An open randomized, prospective, single center; parallel group trial to compare efficiency and safety of PleurX-Pleural Catheter versus standard surgical treatment in patients with malignant pleural effusion and partial entrapment of the lung.

DETAILED DESCRIPTION:
Patients with malignant pleural effusions undergo VATS-procedure. In the intraoperative finding of a partially entrapped lung, patients are randomized in 2 groups.

Arm 1: Insufflation of talc and insertion of a (standard) drainage which will be removed 4-7 days after surgery.

Arm 2: Insufflation of talc and insertion of a (standard) drainage which will be removed 4-7 days after surgery. Additionally, a subcutaneous tunneled catheter will be inserted and will remain in situ

Follow up period is 3 Months

Primary objective is the comparison of quality of life between the 2 arms.

Secondary objective is the reliability of the subcutaneous tunnelled catheter in practice as well as function and dysfunction of the drainage system. Clinical parameters (respiratory function measured as FEV1 and vital capacity, recurrent pleural effusion, infection, need for relief of effusion or pleuracentesis) are observed.

ELIGIBILITY:
Inclusion Criteria:

* One-sided malignant pleural effusion, first occurrence, or following repeated pleuracentesis
* History of dyspnea relieved after pleuracentesis
* Patient is suitable for VATS
* Surgery is indicated by diagnostic necessity
* Ability of subject to understand character and individual consequences of clinical trial
* Written informed consent must be available before enrolment in the trial
* For women with childbearing potential, adequate contraception.
* Histological proven pleural carcinosis by immediate sectioning
* Intraoperative: partial entrapment of the lung

Exclusion Criteria:

* Prior lobectomy or pneumonectomy on the affected side
* The patient is not operable for general reasons or Karnofsky performance score < 50
* Intraoperative suspicion of a pleural empyema
* Chylothorax
* Prior attempts at pleurodesis
* Intended or prior intrapleural chemotherapy or radiotherapy
* Pregnancy and lactation
* Participation in other competing clinical trials and observation period of competing trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
global quality scale QL2 | 3 months

SECONDARY OUTCOMES:
clinical parameters (respiratory function measured as FEV1 and vital capacity, recurrent pleural effusion, infection, need for relief of effusion or pleuracentesis) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hoffmann, MD, PhD, Principal Investigator — Thoraxklinik University of Heidelberg
Locations (1):
- Thoraxklinik, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Putnam JB Jr, Walsh GL, Swisher SG, Roth JA, Suell DM, Vaporciyan AA, Smythe WR, Merriman KW, DeFord LL. Outpatient management of malignant pleural effusion by a chronic indwelling pleural catheter. Ann Thorac Surg. 2000 Feb;69(2):369-75. doi: 10.1016/s0003-4975(99)01482-4. PMID 10735665
- [Background] Tremblay A, Mason C, Michaud G. Use of tunnelled catheters for malignant pleural effusions in patients fit for pleurodesis. Eur Respir J. 2007 Oct;30(4):759-62. doi: 10.1183/09031936.00164706. Epub 2007 Jun 13. PMID 17567670
- [Background] Tremblay A, Michaud G. Single-center experience with 250 tunnelled pleural catheter insertions for malignant pleural effusion. Chest. 2006 Feb;129(2):362-368. doi: 10.1378/chest.129.2.362. PMID 16478853
- [Result] Harzheim D, Sterman D, Shah PL, Eberhardt R, Herth FJ. Bronchoscopic Transparenchymal Nodule Access: Feasibility and Safety in an Endoscopic Unit. Respiration. 2016;91(4):302-6. doi: 10.1159/000445032. Epub 2016 Mar 24. PMID 27007334